CLINICAL TRIAL: NCT06791044
Title: 25(OH)-Vitamin D and Its Association With Bone Density, Body Composition, Strength, Walking Speed, Physical Performance and Pain in Hospitalized Individuals With Neurological Disorders
Brief Title: 25(OH)-Vitamin D and Its Association With Structural and Functional Parameters in Hospitalized Patients With Neurological Diseases
Acronym: NeuroVitD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dionyssiotis, Yannis, M.D. (Individual)
Collaborators: Institute for Rehabilitation and Prevention of Disability Claudius Galenus N.G.O. (Unknown)
Responsible Party: Principal Investigator, Yannis Dionyssiotis, Head of 2nd Physical Medicine and Rehabilitation Department, National Rehabilitation Center EKA, Athens, Greece, Dionyssiotis, Yannis, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFIAPEKA
Record Dates: First submitted 2025-01-12; First posted 2025-01-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Vitamin D Insufficiency
Keywords: 25OHvitD; bone density; body composition; strength; pain; sarcopenia; osteoporosis; sarcopenic obesity; rehabilitation
MeSH Terms: conditions — Pain; Sarcopenia; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vitamin D supplement 1 (Active Comparator): Deltius 50.000 i.u.
  Interventions: Dietary Supplement: DELTIUS
- vitamin D supplement 2 (Active Comparator): Deltius 25.000 I.U. and Deltius 10000 I.U. drops
  Interventions: Dietary Supplement: DELTIUS
- controls (No Intervention): no intervention

INTERVENTIONS:
Dietary Supplement: DELTIUS — A treatment plan will be implemented, as applicable, consisting of 50,000 I.U of vitamin D weekly for 8 weeks
  Arms: vitamin D supplement 1; vitamin D supplement 2
Dietary Supplement: DELTIUS — A treatment plan will be implemented, as applicable, consisting of 25,000 I.U of vitamin D for 4 weeks followed by 10,000 I.U of vitamin D drops weekly for an additional 4 weeks (totaling 8 weeks)
  Arms: vitamin D supplement 1; vitamin D supplement 2

SUMMARY:
The NeuroVitD study aims to assess vitamin D levels in hospitalized cohorts with neurological disorders resulting in motor disabilities, providing epidemiological data necessary for guidelines. The primary objective is to assess vitamin D insufficiency in the neurological populations under investigation and secondary to evaluate the impact of vitamin D supplementation on problems associated with structural and functional parameters.

The NeuroVitD study will be a randomized, cluster, controlled intervention trial lasting 2 years, enrolling 120 individulas, (30 controls), including those with stroke, spinal cord injury, and traumatic brain injury. Comprehensive epidemiological data, including demographic and anthropometric information, will be documented alongside social behaviors such as exercise and smoking. Serum vitamin D levels, bone density, body composition, strength, speed, physical performance and pain will be assessed.

The study will also evaluate the effects of vitamin D supplementation at two distinct dosages: 50,000 I.U of vitamin D weekly for 8 weeks or 25,000 I.U of vitamin D for 4 weeks followed by 10,000 I.U of vitamin D drops weekly for an additional 4 weeks. Calcium, parathyroid hormone, and phosphorus levels will be assessed to examine the impact of vitamin D administration on additional biochemical markers.

The findings will encompass vitamin D levels, bone density, body composition, strength, walking speed, physical performance and pain. The impact of vitamin D supplementation on various biochemical parameters will be analyzed, along with gender and group comparisons. Correlations will be established based on participants' residential locations, the administration of vitamin D supplementation, seasonal variations, and associations with specific medications for neurological conditions.

DETAILED DESCRIPTION:
INTRODUCTION Vitamin D insufficiency in the context of neurodisability has been associated with an elevated risk of poor physical function, bone mineral density and fractures.Clinical experience indicates that the population in Greece generally exhibits lower levels of vitamin D compared to northern European populations. There is a lack of data in Greece concerning persons with neurological motor disorders, and globally, there are no established criteria for vitamin D recommendations.

PURPOSE To assess vitamin D levels in populations with neurological disorders that result in motor disabilities to provide the epidemiological data necessary for the guidelines.

The data from our study will establish a database for any future guidelines regarding vitamin D administration in neurological illnesses, which is now lacking.

The major objective of the study is to determine vitamin D insufficiency in the neurological populations under investigation, while the secondary objective is to assess the impact of vitamin D supplementation on structural and functional parameters.

METHOD The NeuroVitD trial will be a randomized, cluster-based, controlled intervention effectiveness trial of two years. Patient recruitment will occur from June 1, 2025, until June 1, 2027. A total of 120 individuals will participate, with 30 individuals designated as a control group. This includes strokes, spinal cord injuries, traumatic brain injuries, among others.

Comprehensive epidemiological data, including demographic and anthropometric information, along with social habits such as sports participation and smoking, will be documented. Serum vitamin D levels, together with other biochemical markers, bone density, body composition, and metrics of strength, physical performance and speed, if applicable, will be assessed. The assessment will also include safety and tolerance to vitamin D.

Bone density and body composition will be assessed using a DXA machine, strength will be evaluated with a hand dynamometer (utilization contingent upon condition), walking speed will be estimated with the appropriate test, physical performance with SPPB test and pain will be quantified using the proportional pain scale.

Two measurements will be conducted for all parameters, at the commencement and conclusion of the study. New volunteers will be incorporated into the study for a duration of 2 years. The analysis of the results is anticipated in the second half of 2027.

All individuals will be inpatients at the 2nd PMR Department at EKA Hospital and will adhere to the usual rehabilitation procedure tailored to their specific conditions.

Individuals with low vitamin D levels (<20 ng/ml) will be administered a vitamin D supplement, a medically warranted treatment. The control group will consist of individuals with neurological diseases and vitamin D levels exceeding 20 ng/ml.

This study aimed to assess the effects of vitamin D supplementation at two distinct dosages. A treatment plan will be implemented, as applicable, consisting of either 50,000 I.U of vitamin D weekly for 8 weeks or 25,000 I.U of vitamin D for 4 weeks followed by 10,000 I.U of vitamin D drops weekly for an additional 4 weeks (totaling 8 weeks), with an evaluation of which group exhibits superior parameters. The dose that elicits the beneficial impact and is optimal for people with neurological impairment will be assessed. Furthermore, calcium, parathyroid hormone, and phosphorus will be assessed to examine the impact of vitamin D administration on additional biochemical markers.

Exclusion criteria The subject is excluded if they: • are legally or mentally incapable of comprehending and consenting to participate in the study • have a history of or exhibit indicators of metabolic bone disease, including the following: Hypoparathyroidism, primary hyperparathyroidism, recent hyperthyroidism (within the last six months), Paget's disease of bone; no grade 3 or 4 pressure ulcers present; has undergone treatment with pharmacological agents influencing bone metabolism prior to the initial bone density assessment, including the following: Treatment with bisphosphonates in the year prior to the bone density assessment ; Administration of parathyroid hormone in the year prior to the research ; Administration of estrogens, selective estrogen receptor modulators (SERMs), tibolone, or anabolic steroids within the preceding six months. Thyroid drugs are permissible only if the dosage has remained consistent for the preceding six weeks and TSH levels are within the normal range. Corticosteroid medication exceeding 7.5 mg of prednisone orally per day for a duration exceeding one month within the past six months. Immunosuppressant therapy within the past year; Vitamin A therapy above 10,000 IU per day or Vitamin D exceeding 5,000 IU per day. Participants are prohibited from consuming additional vitamin D supplements exceeding 400 IU per day or traveling to regions with heightened sunshine exposure during the trial.

RESULTS The findings will encompass vitamin D levels, bone density, body composition, strength, walking speed and pain. Additionally, the impact of vitamin D supplementation on various biochemical parameters will be analyzed, alongside gender and group comparisons. Correlations will be established based on participants' residential locations (urban or rural), the administration of vitamin D supplementation, seasonal variations, and associations with specific medications for neurological conditions.

Statistical Analysis Our data will be presented using the number of patients (N), mean values (m.s.), and standard deviations for continuous variables, as well as frequencies (n) and percentages (%) for categorical variables. Comparisons of the absolute values of the variables between the two groups (controls vs. neurological lesions) will be conducted using Student's t-test or Welch test (if variances are uneven) and a one-way ANOVA model without repeated measures. For multiple comparisons between time points using pairwise multiple comparison analysis, the investigators will employ the Scheffé test. The General Linear Factorial model will be employed to analyze the factor differences on the measured parameters. Ultimately, the investigators will analyze the differences between the groups by correcting our findings for variables that may influence bone density (such as age and body mass index), employing the general linear factorial model; the tests will be two-sided with a significance threshold of p=0.05. The statistical analysis will utilize the SPSS (Statistical Package for the Social Sciences) software.

The participants will engage in the study following written agreement from themselves or their legal representatives, after being thoroughly informed about the objectives and procedures of the research.

ELIGIBILITY:
Inclusion Criteria:

* populations with neurological disorders
* healthy volunteers (controls)

Exclusion Criteria:

* The subject is excluded if they:

  * are legally or mentally incapable of comprehending and consenting to participate in the study
  * have a history of or exhibit indicators of metabolic bone disease, including the following: Hypoparathyroidism, primary hyperparathyroidism, recent hyperthyroidism (within the last six months), Paget's disease of bone;
  * grade 3 or 4 pressure ulcers present;
  * has undergone treatment with pharmacological agents influencing bone metabolism prior to the initial bone density assessment, including the following: bisphosphonates in the year prior to the bone density assessment ; parathyroid hormone in the year prior to the research ; estrogens, selective estrogen receptor modulators (SERMs), tibolone, or anabolic steroids within the preceding six months.
  * Thyroid drugs are permissible only if the dosage has remained consistent for the preceding six weeks and TSH levels are within the normal range.
  * Corticosteroid medication exceeding 7.5 mg of prednisone orally per day for a duration exceeding one month within the past six months.
  * Immunosuppressant therapy within the past year;
  * Vitamin A therapy above 10,000 IU per day or Vitamin D exceeding 5,000 IU per day.
  * Participants are prohibited from consuming additional vitamin D supplements exceeding 400 IU per day or traveling to regions with heightened sunshine exposure during the trial.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with neurological disease and low levels of vitamin D | up to 12 months
  Number of Participants with neurological diseases eg. stroke, spinal cord injury, traumatic brain injury and low levels of vitamin D

SECONDARY OUTCOMES:
The number of participants with reduced structural and functional parameters due to vitamin D insufficiency and if these parameters are improved with supplements | up to 12 months
  The number of participants with reduced structural and functional parameters due to vitamin D insufficiency and if these parameters are improved with supplements, the impact of vitamin D supplementation on structural parameters eg. bone, body composition and functional parameters eg. muscle strength, walking speed, SPPB test, pain

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Dionyssiotis, Study Chair — National Rehabilitation Center EKA
Locations (2):
- Greece (2):
  - National Rehabilitation Center EKA, Nea Liosia, Athens
  - National Rehabilitation Center EKA (Ethniko Kentro Apokatastasis), Athens, Attica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Di Somma C, Scarano E, Barrea L, Zhukouskaya VV, Savastano S, Mele C, Scacchi M, Aimaretti G, Colao A, Marzullo P. Vitamin D and Neurological Diseases: An Endocrine View. Int J Mol Sci. 2017 Nov 21;18(11):2482. doi: 10.3390/ijms18112482. PMID 29160835
- [Result] Moretti R, Morelli ME, Caruso P. Vitamin D in Neurological Diseases: A Rationale for a Pathogenic Impact. Int J Mol Sci. 2018 Jul 31;19(8):2245. doi: 10.3390/ijms19082245. PMID 30065237
- [Result] Kimball SM, Holick MF. Official recommendations for vitamin D through the life stages in developed countries. Eur J Clin Nutr. 2020 Nov;74(11):1514-1518. doi: 10.1038/s41430-020-00706-3. Epub 2020 Aug 20. PMID 32820241
- Available data/document: Study Protocol — https://eka-hosp.gr/